CLINICAL TRIAL: NCT02609971
Title: Immediate Effects of Whole Body Vibration on Neuromuscular Performance of Quadriceps Femoris in Individuals Submitted to Anterior Cruciate Ligament Reconstruction: A Randomized Clinical Trial
Brief Title: Whole Body Vibration in Individuals Submitted to ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07042915KA
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior cruciate ligament; Neuromuscular Performance and balance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vibration group (Experimental): The vibration group (Vibration at 50 Hz) will hold an exercise protocol on the vibration platform (model Power Plate® pro5 ™), which is to stay on on affected limb, with the knee held in 40 ° of flexion, hands together to the body and the trunk in the erect position. Altogether, the participant will perform 11 sets of 30 seconds with a rest interval of 30 seconds between sets. The knee angle will be monitored throughout the protocol by the second reviewer with a goniometer so that there is no change in it. During the sets the vibrating platform will be turned on at a vibration frequency of 50 Hz.
  Interventions: Other: Vibration at 50 Hz
- Control group (No Intervention): The control group (No vibration) will hold an exercise protocol on the vibration platform, which is to stay on affected limb, with the knee held in 40 ° of flexion, hands together to the body and the trunk in the erect position. Altogether, the participant will perform 11 sets of 30 seconds with a rest interval of 30 seconds between sets. The knee angle will be monitored throughout the protocol by the second reviewer with a goniometer so that there is no change in it. The vibrating platform will remain off throughout intervention.

INTERVENTIONS:
Other: Vibration at 50 Hz — During the exercise protocol, the vibration platform will be turned on at a vibration frequency of 50 Hz.
  Arms: Vibration group

SUMMARY:
The purpose of this study is to analyze the immediate effects of two exercises protocols on the whole body vibration, on the strength of the thigh muscles, joint position sense of the knee and balance in individuals submitted to anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
This is a randomized and blinded clinical trial held at the Laboratory of Neuromuscular Performance of the Department of Physical Therapy, Federal University of Rio Grande do Norte (UFRN). Characterization of the sample: The sample consisted of 46 men submitted to anterior cruciate ligament reconstruction. The participants were randomly divided into 2 distinct groups. Ethical aspects: For its implementation, this project was submitted to the Research Ethics Committee (REC) of the Federal University of Rio Grande do Norte. Was respected and ensured the autonomy and anonymity of participants, as well as privacy as confidential data, as governed Resolution 196/96 of the National Health Council and the Helsinki declaration for human research. Instruments: Stationary bicycle (Ergo-Fit, ErgoCycle 167, Pirmasens, Germany); computerized baropodometry platform Eclipse 3000 model (Guy-Capron® SA, France); vibrating platform model Power Plate® pro5 ™; signal conditioning module (Telemyo direct transmission system) 8-channel (Noraxon, USA); self-adhesive electrode active surface (Noraxon, USA); isokinetic dynamometer (Biodex Multi-Joint System 4, Biomedical Biodex System Inc.®, New York, USA). Procedures: There was a previous pilot study for adequacy of any research procedures and the training of evaluators. The volunteers were informed about the procedures to be performed in the research, signed the informed consent form, fill in an evaluation form with anthropometric data and personal examination of members. Evaluations were performed before and after the intervention protocol. Initially, all the volunteers executed a warming exercise on a stationary bike for 5 minutes. After that, they were submitted for shaving and cleaning the skin with 70% alcohol before attaching the electrodes on vastus medialis and vastus lateralis. Torque rating: the volunteer was positioned sitting on the dynamometer, stabilized by braces and with the device axis aligned with the knee evaluated. The apparatus of the lever arm was attached to the distal leg. Then, it was performed the normalization of the electromyographic signal, where the subject performed two maximal voluntary isometric contractions of knee extension at an angle of 60 ° for 5s, with one-minute interval between each repetition. After, the concentric evaluation was conducted, with 5 maximal contractions for knee flexion and extension at 60 ° / s, starting from 90 ° flexion up to full extension. Joint position sense: The volunteer was instructed to perform a knee extension member starting with 90 ° of flexion. When the 45 target angle wass reached, the dynamometer arm remained in this position, keeping it for 5 seconds, so that the voluntary noticed which the angle to be achieved. Finally, prompted an active extension from 90 ° knee flexion (1 / s) to the target angle, the second trial of the subject. At that moment, the volunteer should trigger a device to record the angle reached. Postural balance: the volunteers were placed standing on the baropodometry platform, supported in the non-dominant member and with the knee kept at 40 ° of flexion. The affected limb remained with the knee in 90 ° of flexion. The evaluation was repeated 3 times, being considered for analysis the average of the two best measures. The evaluation time was 20 seconds on an acquisition frequency of 20 Hz with a period of 1 minute break between tests. Previously the participant was allowed to become familiar with the equipment. Electromyographic activity: emg was collected concurrently with exercise protocols on the platform, as well as during the torque rating.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the 14th and 18th postoperatory week;
* Without pain or inflammatory signs in the joint assessed;
* Absence of labyrinthine and neurological disorders;
* Range of motion greater than 90o flexion and complete extension;
* No previous history of lower limb surgery before the lesion;
* Be performing Physical Therapy

Exclusion Criteria:

* Inability to understand and/or perform the required maneuvers;
* Presence of pain at the time of the tests;
* Complication preventing collection.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Muscle Performance measured through isokinetic dynamometer | Change from baseline in muscle performance at one hour.
  Measured through isokinetic dynamometer. The variable analyzed will be: peak torque normalized by body weight (%).

SECONDARY OUTCOMES:
Muscle activation measured through surface electromyography | Change from baseline in electromyographic activity at one hour.
  Measured by surface electromyography. The variable analyzed will be: RMS (Root Mean Square.